CLINICAL TRIAL: NCT01574534
Title: A Prospective, Randomized, Controlled, Open Label, Multicenter Trial to Test the Non-inferiority of Drug Eluting Balloon vs. Drug Eluting Stent Treatment in de Novo Stenoses of Small Native Vessels Regarding Efficacy and Safety
Brief Title: Basel Stent Kosten Effektivitäts Trial Drug Eluting Balloons vs. Drug Eluting Stents in Small Vessel Interventions
Acronym: BASKET-SMALL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASKET-SMALL2
Record Dates: First submitted 2012-04-08; First posted 2012-04-10 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug eluting balloon (Experimental): paclitaxel-eluting SeQuent® Please balloon, B.Braun Melsungen AG, Berlin, Germany
  Interventions: Device: Drug eluting balloon
- Drug eluting stent (Active Comparator): paclitaxel-eluting Taxus Element® stent, Boston Scientific Corp, Natick MA or everolimus-eluting Xience® stent Abbott Vascular, Santa Clara, California, USA
  Interventions: Device: Drug eluting stent

INTERVENTIONS:
Device: Drug eluting balloon — PCI using paclitaxel-eluting SeQuent® Please balloon, B. Braun Melsungen AG, Berlin, Germany
  Arms: Drug eluting balloon
Device: Drug eluting stent — PCI using paclitaxel-eluting Taxus Element® stent, Boston Scientific Corp, Natick MA
  Arms: Drug eluting stent

SUMMARY:
The investigators hypothesize that in a real-world population undergoing percutaneous coronary intervention (PCI) for de-novo stenoses in small native vessels with a diameter <3 mm, drug eluting balloons (DEB) are non inferior to third-generation drug eluting stents (DES).

DETAILED DESCRIPTION:
Drug-eluting balloons are an established treatment for in-stent stenoses and showed good results in small vessels. Moreover, the available data suggest that DEB are a promising new technique for the treatment of de-novo stenoses in small vessels if pre-dilatation is performed and geographical mismatch is avoided.

The aim of this study is to demonstrate that DEB is non-inferior to DES in a real-world population with respect to the combined clinical endpoint Major adverse cardiac events (MACE), defined as cardiac death, non-fatal myocardial infarction, and target vessel revascularization after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Angina pectoris Canadian Cardiovascular Society (CCS) 2 to 4 or silent ischemia as assessed by stress echocardiography, stress cardiac magnetic resonance, myocardial perfusion scintigraphy, or fractional flow reserve
* PCI of de-novo stenosis in vessels ≥2.0 to <3.0 mm in diameter irrespective of the indication (concomitant PCI of a vessel ≥3.0 mm in diameter is permitted if the stenosis is located in a coronary artery other than the culprit vessel)
* No flow-limiting dissection (TIMI ≤2) or residual stenosis >30% after initial dilatation with a standard or non-compliant balloon, as assessed by the physician in charge
* Written informed consent

Exclusion Criteria:

* Concomitant large-diameter PCI in the same coronary artery (LAD, Ramus circumflexus (RCX), RCA)
* PCI of instent-restenosis (culprit lesion)
* Life expectancy <12 months
* Pregnancy
* Enrolled in another coronary intervention study
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 758 (Actual)
Dates: Start 2012-04; Primary Completion 2018-02-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 12 month
  Major adverse cardiac events (MACE), defined as cardiac death, non-fatal myocardial infarction, and target vessel revascularization after 12 months.

SECONDARY OUTCOMES:
MACE | 24/36 month
  MACE after 24 and 36 months
Revascularization | 12/24/36 month
  The single components of the primary endpoint including target lesion revascularization after 12, 24, and 36 months
Stent Thrombosis | 12/24/36 month
  Possible, probable, and definite stent thrombosis defined according to the ARC criteria after 12, 24, and 36 months; all stent thromboses defined according to the ARC criteria after 12, 24, and 36 months
Thrombolysis In Myocardial Infarction | 12/24/36 month
  Thrombolysis In Myocardial Infarction (TIMI) major bleeding after 12, 24, and 36 months
  Net clinical benefit consisting of the primary endpoint and the TIMI major bleeding after 12, 24, and 36 months
Cost-effectiveness | 12/24/36 month
  Cost-effectiveness of DEB vs. DES after 12, 24, and 36 months
Quantitative Coronary Analysis (QCA) | 12 months
  QCA of patients who had events which required CAG/PCI after Baseline PCI
Outcome in patients with high bleeding risk including patients on OAC | 12 months
  Outcome analyis of patients with high bleeding risk with regard to Major bleeding events (BARC)
Outcome in acute versus stable CAD | 12 months
  Difference of the Population with acute versus stable CAD with regard to baseline characteristics, primary and secondary outcome measures (MACE, stent thrombosis, major bleeding)
Outcome in diabetics vs non diabetics | 12 months
  Difference of the diabetic versus non-diabetic population regarding baseline characteristics and primary and secondary outcome measures (MACE, stent thrombosis, major bleeding)
sex specific inequalities in the use of drug coated balloons for small coronary artery disease | 12 months
  sex specific difference in baseline charchteristics, Impact of sex on safety and efficacy in the stent-free strategy regarding primary and secondary endpoint (MACE, stent thrombosis, major bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Raban V Jeger, PD Dr, Principal Investigator — Cardiology, University Hospital Basel
Locations (14):
- Medizinische Universität Graz Kardiologie, Graz, Austria
- Germany (9):
  - Cardiology, Zentralklinik Bad Berka, Bad Berka
  - Unfallkrankenhaus Berlin, Dept. Internal Medicine, Berlin
  - Charité Universitätsmedizin Berlin, Kardiologie, Berlin
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau
  - Klinikum Westfalen GmbH Knappschaftskrankenhaus, Dortmund
  - Universitätsklinikum des Saarlandes - Kardiologie, Angiologie und internistische Intensivmedizin, Homburg/Saar
  - University Hospital Jena, Jena
  - Herzzentrum Leipzig GmbH, Universitätsklinik, Leipzig
  - Department of Internal Medicine/Cardiology, University Hospital Ulm, Ulm
- Switzerland (4):
  - Cardiology, University Hospital Basel, Basel
  - Cardiology Cantonal Hospital Baselland Liestal, Liestal
  - Luzerner Kantonsspital, Lucerne
  - Cardiology, Kantonsspital St. Gallen, Sankt Gallen

REFERENCES:
- [Background] Gilgen N, Farah A, Scheller B, Ohlow MA, Mangner N, Weilenmann D, Wohrle J, Jamshidi P, Leibundgut G, Mobius-Winkler S, Zweiker R, Krackhardt F, Butter C, Bruch L, Kaiser C, Hoffmann A, Rickenbacher P, Mueller C, Stephan FP, Coslovsky M, Jeger R; BASKET-SMALL 2 Investigators. Drug-coated balloons for de novo lesions in small coronary arteries: rationale and design of BASKET-SMALL 2. Clin Cardiol. 2018 May;41(5):569-575. doi: 10.1002/clc.22942. Epub 2018 May 10. PMID 29527709
- [Result] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Derived] Rubini Gimenez M, Scheller B, Farah A, Ohlow MA, Mangner N, Weilenmann D, Wohrle J, Cuculi F, Leibundgut G, Mobius-Winkler S, Cattaneo M, Gilgen N, Kaiser C, Jeger RV. Sex-specific inequalities in the use of drug-coated balloons for small coronary artery disease: a report from the BASKET-SMALL 2 trial. Clin Res Cardiol. 2024 Jul;113(7):959-966. doi: 10.1007/s00392-023-02249-6. Epub 2023 Jul 26. PMID 37495797
- [Derived] Scheller B, Rissanen TT, Farah A, Ohlow MA, Mangner N, Wohrle J, Mobius-Winkler S, Weilenmann D, Leibundgut G, Cuculi F, Gilgen N, Coslovsky M, Mahfoud F, Jeger RV; BASKET-SMALL 2 Investigators. Drug-Coated Balloon for Small Coronary Artery Disease in Patients With and Without High-Bleeding Risk in the BASKET-SMALL 2 Trial. Circ Cardiovasc Interv. 2022 Apr;15(4):e011569. doi: 10.1161/CIRCINTERVENTIONS.121.011569. Epub 2022 Apr 12. PMID 35411792
- [Derived] Mangner N, Farah A, Ohlow MA, Mobius-Winkler S, Weilenmann D, Wohrle J, Linke A, Stachel G, Markovic S, Leibundgut G, Rickenbacher P, Cattaneo M, Gilgen N, Kaiser C, Scheller B, Jeger RV; BASKET-SMALL 2 Investigators. Safety and Efficacy of Drug-Coated Balloons Versus Drug-Eluting Stents in Acute Coronary Syndromes: A Prespecified Analysis of BASKET-SMALL 2. Circ Cardiovasc Interv. 2022 Feb;15(2):e011325. doi: 10.1161/CIRCINTERVENTIONS.121.011325. Epub 2022 Jan 10. PMID 35000455
- [Derived] Wohrle J, Scheller B, Seeger J, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Weilenmann D, Stachel G, Leibundgut G, Rickenbacher P, Cattaneo M, Gilgen N, Kaiser C, Jeger RV; BASKET-SMALL 2 Investigators. Impact of Diabetes on Outcome With Drug-Coated Balloons Versus Drug-Eluting Stents: The BASKET-SMALL 2 Trial. JACC Cardiovasc Interv. 2021 Aug 23;14(16):1789-1798. doi: 10.1016/j.jcin.2021.06.025. PMID 34412797
- [Derived] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Weilenmann D, Wohrle J, Stachel G, Markovic S, Leibundgut G, Rickenbacher P, Osswald S, Cattaneo M, Gilgen N, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Long-term efficacy and safety of drug-coated balloons versus drug-eluting stents for small coronary artery disease (BASKET-SMALL 2): 3-year follow-up of a randomised, non-inferiority trial. Lancet. 2020 Nov 7;396(10261):1504-1510. doi: 10.1016/S0140-6736(20)32173-5. Epub 2020 Oct 19. PMID 33091360
- [Derived] Fahrni G, Scheller B, Coslovsky M, Gilgen N, Farah A, Ohlow MA, Mangner N, Weilenmann D, Wohrle J, Cuculi F, Leibundgut G, Mobius-Winkler S, Zweiker R, Twerenbold R, Kaiser C, Jeger R; BASKET-SMALL 2 Investigators. Drug-coated balloon versus drug-eluting stent in small coronary artery lesions: angiographic analysis from the BASKET-SMALL 2 trial. Clin Res Cardiol. 2020 Sep;109(9):1114-1124. doi: 10.1007/s00392-020-01603-2. Epub 2020 Jan 29. PMID 31993736